CLINICAL TRIAL: NCT06666049
Title: Gastric POCUS for Airway Management in Patients Using Glucagon-like Peptide-1 Receptor Agonist
Acronym: POCUS
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: POCUS
Record Dates: First submitted 2024-10-22; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Aspiration Pneumonia
Keywords: Bronchopulmonary complications; Ultrasound
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment with GLP-1 agonists: Patients undergoing treatment with GLP-1 agonists, from any geographical area, who choose to undergo scheduled and/or urgent surgery under general anesthesia and/or sedation at our hospital over a two-year period (2024-2025).
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — Gastric Ultrasound

SUMMARY:
1. Introduction

Scheduled surgery requires patients to undergo a preoperative fasting period of at least 6 hours to ensure an empty stomach, significantly reducing the risk of perioperative aspiration pneumonia. However, certain medications and/or conditions have been described that can cause delayed gastric emptying, potentially placing patients at risk for aspiration; among these entities are diabetic gastroparesis and the use of GLP-1 analogs as a treatment for diabetes.

Glucagon-like peptide-1 (GLP-1) is an intestinal hormone with beneficial effects on blood glucose control. It stimulates insulin release, reduces glucagon production, and decreases appetite, making it a therapeutic tool for the treatment of type 2 diabetes and obesity. GLP-1 receptor agonists have been approved by the FDA for these indications, and their use is continuously increasing. One of the primary side effects of GLP-1 agonists is delayed gastric emptying, which can lead to nausea, vomiting, and abdominal distension. Recent scientific literature has presented multiple reports demonstrating delayed gastric emptying associated with the use of GLP-1 agonists, including cases of pulmonary aspiration during anesthesia (despite adequate fasting periods). These findings underscore the necessity for anesthesiologists and perioperative physicians to be aware of the potential risks associated with these medications. It is suggested that these drugs be discontinued days prior to elective surgical procedures, depending on dosing frequency. It is essential to assess the presence of gastrointestinal symptoms, as they may indicate an increase in residual gastric content and heighten the risk of complications. As the use of GLP-1 agonists continues to expand, it is crucial to recognize and manage the risks associated with delayed gastric emptying in patients utilizing these agents. Further research is needed to establish more precise guidelines and mitigate the perioperative risks associated with these drugs.

DETAILED DESCRIPTION:
2. Hypothesis

The study will be based on two working hypotheses:

Gastric ultrasonography performed by trained anesthesiologists is a useful tool for assessing gastric content and making clinical decisions regarding airway management.

3. Methodology

The reference population will consist of patients undergoing scheduled surgery with a conventional preoperative fasting period (at least 6 hours).

Inclusion criteria for the study will be:

Patients taking GLP-1 analog medications. Adults over 18 years of age. Patients undergoing scheduled surgery after a fasting period greater than 6 hours and less than 8 hours (first patient of the morning surgical schedule).

Patients who have been properly informed and have signed the informed consent form, expressing their agreement to participate in the study.

ASA I-III classification. Sufficient intellectual capacity to understand the procedure and the equipment used.

Exclusion criteria will include:

Not meeting the previously stated criteria. History of esophagogastric pathology or previous abdominal surgery. Hiatal hernia/gastroesophageal reflux disease. Autonomic nervous system disorders. Neurological or neuromuscular diseases. Use of medications/drugs that affect autonomic regulation and delay gastric emptying (opioids) or potentiate it (prokinetics).

Pregnancy. Presence of arrhythmias.

4. Description of the Intervention

Immediately prior to surgery, a gastric ultrasound will be performed on the patient in both supine and right lateral decubitus positions. A qualitative, semi-quantitative, and quantitative measurement of gastric content and volumes will be conducted according to the algorithm designed by Perlas et al. Data will be recorded in the researcher's data collection notebook. Following this, the anesthetic and surgical procedures will proceed as planned.

5. Ethical, Legal, and Economic Considerations

Patients who choose to participate in the study will be asked for both verbal and written consent (see patient information sheet and informed consent form). Since the study is purely observational and will involve no interventions, there will be no legal liability arising from the study that necessitates insurance coverage. Any ultrasound machine available in the anesthesia department will be used for the study, meaning that conducting the study will not incur any additional costs for the hospital.

6. Results

The results will be analyzed by the study investigators, with the ultimate goal of publication in a relevant specialty journal. If any results are applicable for improving standard clinical practice in our hospital, they will be communicated to the Department of Anesthesiology and Resuscitation and to any other interested parties through a clinical session.

ELIGIBILITY:
Inclusion Criteria:

Adults patients ,ASA I-III, taking GLP-1 analog medications, undergoing scheduled surgery.

Exclusion Criteria:

1. - History of esophagogastric pathology or previous abdominal surgery.
2. - Hiatal hernia/gastroesophageal reflux disease.
3. - Autonomic nervous system disorders.
4. - Neurological or neuromuscular diseases.
5. - Use of medications/drugs that affect autonomic regulation and delay gastric emptying (opioids) or potentiate it (prokinetics).
6. - Pregnancy.
7. - Presence of arrhythmias.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The reference population will consist of patients undergoing scheduled surgery with a conventional preoperative fasting period (at least 6 hours).
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Gastric Ultrasound | 5 minutes
  Gastric ultrasonography performed by trained anesthesiologists, for measuring gastric content in volume (cm3) is a useful tool for assessing gastric content and making clinical decisions regarding airway management.

SECONDARY OUTCOMES:
weight in kilograms | 1 minute
  Weight in kilograms
Height in centimeters | 1 minute
  Height in centimeters
BMI in kg/m^2 | 1 minute
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad Navarra, Madrid, Spain